CLINICAL TRIAL: NCT00005874
Title: Phase II Study of RFS 2000 (9-Nitro-Camptothecin, 9-NC) in Patients With Soft-Tissue Sarcomas
Brief Title: Nitrocamptothecin in Treating Patients With Soft Tissue Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067910; SUPERGEN-RFS2000-24; MDA-DM-99109
Record Dates: First submitted 2000-06-02; First posted 2004-04-13 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-09

CONDITIONS: Gastrointestinal Stromal Tumor; Sarcoma; Small Intestine Cancer
Keywords: adult leiomyosarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; small intestine leiomyosarcoma; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; childhood leiomyosarcoma; gastrointestinal stromal tumor; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma; Leiomyosarcoma | interventions — rubitecan

INTERVENTIONS:
Drug: rubitecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of nitrocamptothecin in treating patients who have locally advanced or metastatic soft tissue sarcomas.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy and toxicity of nitrocamptothecin in patients with locally advanced or metastatic gastrointestinal leiomyosarcomas or other soft tissue sarcomas.

OUTLINE: Patients are stratified by disease (gastrointestinal leiomyosarcomas vs other soft tissue sarcomas). Patients receive oral nitrocamptothecin daily on days 1-5. Treatment continues weekly in the absence of disease progression or unacceptable toxicity. Responding patients who undergo surgery then receive an additional 4-6 courses (4 weeks/course).

PROJECTED ACCRUAL: A total of 34-78 patients (17-39 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed locally advanced or metastatic inoperable soft tissue sarcoma Measurable or evaluable disease that has not been irradiated Must have received, refused, or be not eligible for doxorubicin/ifosfamide treatment Previously untreated gastrointestinal leiomyosarcoma allowed

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 3 times normal Renal: Creatinine less than 2.0 mg/dL Cardiovascular: No New York Heart Association class III or IV heart disease No active coronary disease requiring therapy Pulmonary: No severe pulmonary insufficiency Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study No other prior malignancy in past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix No concurrent active infections No psychosis or mental disability that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 7 days since prior biological therapy and recovered No concurrent immunotherapy Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy and recovered No other concurrent chemotherapy Endocrine therapy: At least 7 days since prior hormonal therapy and recovered Radiotherapy: See Disease Characteristics Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-06; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Show-Li Sun, MD, Study Chair — Astex Pharmaceuticals, Inc.
Locations (1):
- SuperGen, Incorporated, Dublin, California, United States